CLINICAL TRIAL: NCT05393297
Title: InGReS: Intra-treatment Image Guided Adaptive Radiotherapy Dose-escalation Study
Acronym: InGReS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Teresa Guerrero Urbano, Consultant Clinical Oncologist, Guy's and St Thomas' NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22/LO/0056; 257601 (Other: IRAS)
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Cancer
Keywords: Radiotherapy; Adaptive; Dose-escalation; Oropharyngeal Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HNSCC receiving (chemo)radiotherapy (Experimental): Radiation: Intra-treatment FDG-PET-CT and MRI will be used to identify tumours and patients for dose-escalation. Patients identified for dose-escalation (boost) will undergo adaptive radiotherapy replanning, with the primary tumour (GTVp) receiving 76.9Gy in 35 fractions.
  Interventions: Diagnostic Test: Imaging: Intra-treatment FDG-PET-CT and MRI; Radiation: Intra-treatment Image-Guided Adaptive Radiotherapy Dose-escalation

INTERVENTIONS:
Diagnostic Test: Imaging: Intra-treatment FDG-PET-CT and MRI — FDG-PET-CT and MRI scan will be used during radiotherapy to assess early treatment response and identify tumours eligible for dose-escalation.
Radiation: Intra-treatment Image-Guided Adaptive Radiotherapy Dose-escalation — Tumours eligible for dose-escalation (boost), as seen on intra-treatment FDG-PET-CT and MRI scan, will receive 76.9 Gy to the residual gross primary tumour. The radiotherapy plan will be replanned to incorporate the simultaneous-integrated-boost to the GTVp which will be delivered over the last 3 weeks of treatment

SUMMARY:
InGReS is a phase I pilot study of adaptive dose-escalated radiotherapy in combination with platinum-based chemotherapy (CRT) for locally advanced head and neck cancer.

InGReS will assess the feasibility of adapting the radiotherapy (RT) plan for each patient, based on anatomical and metabolic changes in the tumour seen on MRI and FDG-PET-CT performed after 2 weeks of CRT in a multicentre setting. The overall aim of the trial is to determine the safety and feasibility of delivering dose-escalated Intensity Modulated Radiotherapy (IMRT) to the residual primary tumour, as seen on intra-treatment imaging, in the final 3 weeks of RT.

DETAILED DESCRIPTION:
The study will recruit 15 patients with locally advanced oropharyngeal or hypopharyngeal squamous cell carcinoma (SCC) who are suitable for primary treatment with concurrent chemo-radiation. The main aim is to see whether it is feasible to perform a FDG positron emission tomography-computed tomography (FDG-PET-CT) and Magnetic Resonance Imaging (MRI) scan after 2 weeks of radiotherapy and re-plan the radiotherapy to escalate the dose of radiotherapy delivered to the residual primary tumour as seen on PET-CT and MRI.

Patients will commence with standard chemo-radiotherapy; 70 Gray (Gy) in 35 fractions with concomitant platinum chemotherapy. After 2 weeks of chemo-radiotherapy patients will have an intra-treatment FDG-PET-CT and MRI scan to assess early response to treatment. Patients with evidence of residual disease will proceed with the dose-escalation phase of the study, with an adaptive radiotherapy re-plan and dose-escalation to the residual primary tumour.

The study will establish acute and late radiotherapy toxicity rates in patients who receive dose-escalated RT, particularly the effect of treatment on long-term swallowing function. The study hypothesis is that mucosal toxicity rates for dose-escalated treatment will be equivalent to those for standard CRT, according to published data. Furthermore, it will also explore whether changes in FDG-PET-CT and MRI during treatment correlate with patient outcomes and potential blood-based biomarkers of treatment response. Local control, disease-free and overall survival will be assessed for both standard and dose-escalated approaches.

ELIGIBILITY:
Inclusion criteria:

1. Locally advanced, histologically confirmed squamous cell carcinoma (SCC) of the oropharynx and hypopharynx to be treated with primary radical chemo-radiotherapy:

   1. Hypopharyngeal cancer - HPV negative OR HPV positive
   2. Oropharyngeal cancer - EITHER HPV negative OR HPV positive with N stage at least N2b and greater than 10 pack year smoking history: All HPV positive oropharyngeal patients should have at least stage III disease (TNM8)
2. ≥T2 tumours:
3. Staging MRI showing minimum diameter of primary tumour greater than or equal to 1cm
4. Staging 18F-FDG-PET/CT showing adequate uptake in the primary tumour, defined as SUVmax of ≥ 5.0
5. Multidisciplinary team (MDT) decision to treat with primary CRT with curative intent
6. Patients fit for radical treatment with primary CRT
7. WHO Performance Status 0-1

Exclusion criteria:

1. Previous radiotherapy to the head and neck region interfering with the protocol treatment plan
2. Patients requiring neo-adjuvant chemotherapy
3. Inability to tolerate PET or MRI; general contra-indications to MRI
4. Contra-indication to gadolinium
5. Baseline SUVmax < 5.0 in the primary tumour on PET-CT or smaller than 1cm in axial dimensions on cross sectional imaging
6. GFR <40ml/min
7. Previous primary malignancy within 2 years (excluding adequately treated non-melanoma skin cancer, low risk Prostate cancer Gleason 6 or below, carcinoma in situ of cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-06-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of delivering an additional 10% dose (biological rather than numerical) of radiotherapy to the residual primary tumour during radiotherapy | 12 months
  Incidence of grade 3 or above late Radiation Therapy Oncology Group (RTOG) and European Organization for Research and Treatment of Cancer (EORTC) mucosal toxicity or feeding tube retention rate following completion of treatment. An excess rate of >14% would be regarded as unacceptable.

SECONDARY OUTCOMES:
Incidence of grade 4 acute mucosal toxicity (NCI CTCAE) | 12 weeks
  Toxicity grading, using National Cancer Institute Common Terminology Criteria for Adverse Events scale v.5.0, will be presented during and up to 12 weeks after treatment. Grading scale: 0-5, with the higher score meaning a worse outcome.
Incidence of grade 3 or above late non-mucosal toxicity (NCI CTCAE) | 12 months
  Toxicity of non-mucosal late toxicity will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events scale v.5.0. Scores will be presented at 13 weeks; 6 and 12 months after treatment. Grading scale: 0-5, with the higher score meaning a worse outcome.
Incidence of grade 3 or above late non-mucosal toxicity (RTOG/EORTC) | 12 months
  Toxicity of non-mucosal late toxicity will be graded using Radiation Therapy Oncology Group (RTOG) and European Organization for Research and Treatment of Cancer (EORTC) late toxicity scoring. Scores will be presented at 13 weeks; 6 and 12 months after treatment. Grading scale: 0-5, with the higher score meaning a worse outcome.
Incidence of grade 3 or above late non-mucosal toxicity (LENT/SOMA criteria) | 12 months
  Toxicity of non-mucosal late toxicity will be graded using the modified Late Effects on Normal Tissues- Subjective, Objective, Management, Analytic (LENTSOMA) scoring systems. Scores will be presented at 13 weeks; 6 and 12 months after treatment. Grading scale: 0-4, with the higher score meaning a worse outcome.
To assess swallowing panel measurements including qualitative swallowing assessments (MDADI) | 12 months
  M.D. Anderson Dysphagia Inventory (MDADI) scores will be plotted over time. Scores will be presented at baseline and weeks 3 & 7 of CRT. Then at 13 weeks; 6 and 12 months after treatment. A higher MDADI score represents better function and quality of life.
To assess patient reported outcomes measures and quality of life questionnaires (UW-QOL v 4.1) | 12 months
  Patient reported outcomes measures and quality of life scores using the University of Washington Quality of Life Questionnaire (UW-QOL) v4.1 will be plotted over time. Scores will be presented at baseline and weeks 3 & 7 of CRT. Then at 13 weeks; 6 and 12 months after treatment. A higher score represents better function and quality of life.
To assess patient reported outcomes measures and quality of life questionnaires (EORTC QLQ-C30 and EORTC QLQ-H&N43) | 12 months
  Patient reported outcomes measures and quality of life scores, using the questionnaires of the European Organisation for Research and Treatment of Cancer Head and Neck Cancer Modules 30 and 43 (EORTC QLQ-C30 and EORTC QLQ-H&N43), will be plotted over time. Scores will be presented at baseline and weeks 3 & 7 of CRT. Then at 13 weeks; 6 and 12 months after treatment.
  For the functioning and the quality of life scales, a higher score indicates better health. For the symptoms scales, a higher score indicates a higher level of symptom burden.
To assess results of quantitative swallowing assessments (Videofluoroscopy) | 12 months
  Video-fluoroscopy test scores, particularly the Rosenbek Penetration/Aspiration Scale (PAS) and the summary Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) scores, will be presented at 12 months after treatment. For both PAS and summary DIGEST scores, a higher score indicates worse function.
To assess late toxicity rates and the effect of treatment on swallowing function (100ml water swallow) | 12 months
  100ml water swallow test results will be presented at baseline. Then at 6 weeks, 13 weeks, 6 months and 12 months after treatment. Patients will be reported as having failed the test if they coughed or had a wet voice quality post swallow or were unable to finish the task.
To assess tumour response to adaptive radiotherapy dose-escalation (FDG-PET-CT) | 3 months
  Complete metabolic response rate on PET-CT scan will be reported at 3 months after treatment
The loco-regional tumour control | 12 months
  Incidence of local or regional tumour recurrence rates will be presented.
Disease-free survival | 12 months
  Disease-free survival rates (Kaplan-Meier estimates) will be presented at 3 and 12 months after completion of CRT.
Overall survival | 12 months
  Overall survival rates (Kaplan-Meier estimates) will be presented at 3 and 12 months after completion of CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Guerrero Urbano, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No